CLINICAL TRIAL: NCT04904705
Title: The Effect of the Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach for Children With Organic Acidemia on Daily Life Activities, Quality of Life and Participation
Brief Title: The Effect of the Cognitive Orientation to Daily Occupational Performance Approach for Children With Organic Acidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Leman Dursun, Occupational Therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA-20057
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Organic Acidemia; Cognitive Orientation
Keywords: Organic Acidemia; Cognitive Orientation; Activities of Daily Living; Participation; Quality of Life; Telerehabilitation
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: In consequence of the statistical power analysis, the number of individuals to participate in the study was determined as 34 children diagnosed with organic acidemia, including 17 in the intervention group and 17 in the control group. The study will be conducted in a randomized controlled method. Children will be divided into intervention and control groups by using a computer-assisted online randomization application. Participants will be randomly numbered and randomly assigned to the intervention or control group without repeating the same number with the online randomization application available at randomizer.org. Both groups will be given a home program that will be prepared and sent to the person via e-mail. The Cognitive Orientation for Daily Occupational Performance (CO-OP) Approach to the intervention group will be applied by video conferencing method in a total of 10 sessions, 2 sessions per week, through 5 weeks, and a total of 12 sessions with initial and final evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach (Active Comparator): It will be given a home program. Then The Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach will be applied by video conferencing method in a total of 10 sessions, 2 sessions per week, through 5 weeks, and a total of 12 sessions with initial and final evaluations.
  The Cognitive Orientation for Daily Activity Performance (CO-OP) approach is a person-oriented, performance-solving. and problem-solving approach that enables strategy acquisition and guided exploration for the acquisition and learning of new skills.
  Interventions: Other: The Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach; Other: Home Program
- Home Program (Active Comparator): It will be given a home program only.
  Interventions: Other: Home Program

INTERVENTIONS:
Other: The Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach — The Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach is a cognitive-based approach. This is a person-oriented, performance-solving problem-solving approach that enables strategy acquisition and guided exploration for the acquisition and learning of new skills.
  The main objectives of this approach are; define and transfer domain-specific strategies to other motor-based tasks to gain skills, learn problem-solving strategy (goal, plan, do, check) and adapt to other environments (such as home, school).
  Arms: Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach
Other: Home Program — Home Program are activities that a participant can apply at home to improve their skills.

SUMMARY:
The aim of this study is to research the effect of Cognitive Orientation to daily Occupational Performance (the CO-OP Approach) on daily life activities, quality of life and participation in children with organic acidemia.

The hypotheses of the study are as follows:

* Cognitive Orientation to daily Occupational Performance (the CO-OP Approach) applied to children with organic acidemia has no effect on daily life activities.
* Cognitive Orientation to daily Occupational Performance (the CO-OP Approach) applied to children with organic acidemia has no effect on quality of life.
* Cognitive Orientation to daily Occupational Performance (the CO-OP Approach) applied to children with organic acidemia has no effect on participation.

DETAILED DESCRIPTION:
Organic acidemia is an inherited metabolic diseases due to the deficiency of an enzyme or a transport protein involved in one of the several cellular metabolic pathways devoted to the catabolism of amino acids, carbohydrates, or lipids. Collectively, their incidence approximates 1 out of 3000 live births. Moreover, the demanding medical management of organic acidemia patients often dominates the efforts of their metabolic teams, impacting on time dedicated toward addressing aspects of care that could enhance functional independence and improve quality of life. While most published data on long-term organic acidemia outcomes have focused on medical endpoints such as survival and neurocognition, there have been fewer efforts to document functionality, independence, and social integration or the need for rehabilitation interventions that could maintain and maximize function. It's understood that delivering one form of meta-cognitive strategy training, the CO-OP approach, using a telerehabilitation format is feasible and shows similar positive effects to face-to-face delivery.

It was planned to include children between the ages of 7-12 who were diagnosed with organic acidemia in this study. In consequence of the statistical power analysis, the number of individuals to participate in the study was determined as 34 children diagnosed with organic acidemia, including 17 in the intervention group and 17 in the control group. The study will be conducted in a randomized controlled method. Children will be divided into intervention and control groups by using a computer-assisted online randomization application that provides an equal number and probability. Participants will be randomly numbered and randomly assigned to the intervention or control group without repeating the same number with the online randomization application available at randomizer.org. Both groups will be given a home program. Home programs will be prepared and sent to the person via e-mail. The Cognitive Orientation for Daily Activity Performance (CO-OP) Approach to the intervention group will be applied by video conferencing method in a total of 10 sessions, 2 sessions per week, through 5 weeks, and a total of 12 sessions with initial and final evaluations.

The children to be included in our study will be determined among the children with organic acidemia who are directed from Hacettepe University Metabolism and Nutrition Department. The contact information of the volunteers who agree to participate in the study will be given to the occupational therapist. The occupational therapist will provide information on how to download and use the video interview program called Zoom on his/her phone or computer. The session schedule will be determined after the program is set up. The program named Zoom was preferred because it is free, easy to install, and accessible compared to the other video conference programs.

The informed consent form will be sent to the individuals online by using Google Forms. After the participants approve the consent form, they will reach the evaluations to be prepared on Google Forms. One of the evaluation scales, the Canadian Occupational Performance Measure (COPM) will be made over the video interview. If they do not want to approve the consent form, they will be exempted from the study by checking the "I do not approve" option.

In this study, Canadian Occupational Performance Measure (COPM), Pediatric Evaluation of Disability Inventory (PEDI), The Child and Adolescent Scale of Participation (CASP), Quality of Life Questionnaire for Children (Kid-KINDL), Assistance to Participate Scale, and Sociodemographic Questionnaire will be implemented.

ELIGIBILITY:
Inclusion criteria:

* Children between the ages of 7-12
* Being diagnosed with organic acidemia
* Being able to read and write
* Having sufficient language skills to be able to communicate and be understood during the intervention

Exclusion criteria:

* Being on other treatment
* Having significant vision or hearing problems
* Refusing to participate in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | In the first week and the sixth week
  The Canadian Occupational Performance Measure (COPM) is designed to be used for client-centred clinical practice. The COPM is an outcome measure designed for use by occupational therapists to assess client outcomes in the areas of self-care, productivity and leisure. Using a semi-structured interview, the COPM is a five step process which measures individual, client-identified problem areas in daily function. Two scores, for performance and satisfaction with performance are obtained.
Quality of Life Questionnaire for Children (Kid-KINDL) | In the first week and the sixth week
  The Kid-KINDL questionnaire contains 6 dimensions (viz, physical well-being, emotional well-being, self-esteem, friends, family, and school), each of them including 4 items. Each item in the test is 5-point Likert-scaled (positively worded items: never scores 1 and always scores 5; negatively worded items: never scores 5 and always scores 1). 7 From the item scores, the total Kid-KINDL score and each dimension score can be calculated and transformed into a 0 to 100 result.
The Child and Adolescent Scale of Participation (CASP) | In the first week and the sixth week
  The CASP specifically measures children's extent of participation and restrictions in home, school and community life situations and activities compared to same-age peers as reported by family caregivers. It consists of 20 items divided into four sub-sections: (1) Home Participation, (2) School Participation, (3) Community Participation and (4) Home and Community Living Activities. Each item addresses a broad participation domain with examples provided for each domain (see Appendix for item descriptions). The 20 items are rated on a 4-point scale (4 = Age expected, 3 = Somewhat restricted, 2 = Very restricted, 1 = Unable) or as 'Not applicable'.
Pediatric Evaluation of Disability Inventory (PEDI) | In the first week and the sixth week
  The Pediatric Evaluation of Disability Inventory (PEDI) is a comprehensive functional assessment designed for use by physical and occupational therapists, as well as other rehabilitation and educational professionals. The PEDI measures both functional performance and capability in three domains: (1) self-care, (2) mobility, and (3) social function. The PEDI consists of 197 functional skill items, and 20 items that assess caregiver assistance and modifications.
Assistance to Participate Scale (APS) | In the first week and the sixth week
  Assistance to Participate Scale (APS) measures the level of assistance that a school-aged child with a disability needs to participate in game, leisure, and recreational activities at home and in the community, from the perspective of the primary caregiver. It takes 5-10 min to answer the APS by the caregivers. Participants were asked to rate the level of assistance that they typically provide to their child on a 5-point ordinal scale (1 = Unable to participate; 2 = Participates with my assistance at all stages of the activity; 3 = Participates after I have set him/her up and help at times during the activity; 4 = Participates with my supervision only; 5 = Participates independently). The minimum and maximum scores range between 8 and 40. Lower scores indicate requirement of higher levels of assistance.
Sociodemographic Questionnaire | In the first week
  Data on gender, age, height, weight, dominant hand, school class, medicine names used before will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Ph.D., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No